CLINICAL TRIAL: NCT02187029
Title: A Randomized, Double Blind, Third Party Open, Placebo Controlled Multi-center Study Of Efficacy, Safety And Tolerability Of Pf-06743649 In Gout Subjects
Brief Title: Efficacy, Safety And Tolerability Of PF-06743649 In Gout Subjects.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: B7911002 was prematurely discontinued due to a safety concern that led to decision to terminate the study on 10 Nov 2014
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B7911002
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-09

CONDITIONS: Gout
Keywords: Hyperuricemia; gout; serum uric acid
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-06743649 dose level 1 (Cohort 1) (Experimental)
  Interventions: Drug: PF-06743649
- Placebo for PF-06743649 (Cohort 1) (Placebo Comparator)
  Interventions: Other: Placebo
- PF-06743649 dose level 2 (Cohort 2) (Experimental)
  Interventions: Drug: PF-06743649
- Placebo for PF-06743649 (Cohort 2) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-06743649 — Daily dosing (dose level 1) tablet for 14 days
  Arms: PF-06743649 dose level 1 (Cohort 1)
Other: Placebo — Daily dosing (tablet) for 14 days
  Arms: Placebo for PF-06743649 (Cohort 1)
Drug: PF-06743649 — Daily dosing (dose level 2) tablet(s) for 14 days
  Arms: PF-06743649 dose level 2 (Cohort 2)
Other: Placebo — Daily dosing (tablets) for 14 days
  Arms: Placebo for PF-06743649 (Cohort 2)

SUMMARY:
The purpose of the study is to assess the effect of PF-06743649 in lowering serum uric acid in subjects suffering from gout following 14 days of dosing, as well as assessing safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets the diagnosis of gout as per the American Rheumatism Association Criteria for the Classification of acute Arthritis of Primary Gout.
* Subjects taking urate lowering therapy at the time of screening must be willing to discontinue their prior urate lowering therapy from the time of Screening Visit 1 until completion of the study period Day 16.
* Subjects taking urate lowering therapy at the time of screening must have a serum urate level of >= 8.0 mg/dL at time of the second screening visit.
* Subjects NOT taking urate lowering therapy at the time of screening must have a serum urate level of >= 8.0 mg/dL at both screening visits 1 and 2.

Exclusion Criteria:

* Positive medical history or current evidence of medical or psychiatric condition/disease, or ECG or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
* Chronic kidney disease classified as moderate or severe (Clinical Practice Guideline, National Kidney Foundation)12; with GFR < 60 mL/min/1.73m2 calculated by the Cockcroft-Gault equation.
* Subjects with current tophaceous gout.
* Gout flare that has not resolved for at least 2 weeks prior to randomization.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - MRA Clinical Research, LLC, Miami, Florida
  - Miami Research Associates, Inc., South Miami, Florida
  - Vince and Associates Clinical Research Inc., Overland Park, Kansas
  - Vince and Associates Clinical Research, Inc., Overland Park, Kansas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7911002&StudyName=Efficacy%2C%20Safety%20And%20Tolerability%20Of%20PF-06743649%20In%20Gout%20Subjects.%0A

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: PF-06743649 2.5 mg to 10 mg: Following a dose titration regimen, participants received PF-06743649 2.5 mg tablet orally once daily (QD) for 8 days, followed by PF-06743649 10 mg QD for 6 days.
- Cohort 1: PF-06743649 40 mg: Prior to dose titration, participants received PF-06743649 40 mg tablet orally QD for 14 days.
- Cohort 2: PF-06743649 5 mg: Participants received PF-06743649 5 mg tablets QD for 2 days before the study was terminated for safety reasons. This cohort was stopped after acute kidney injury was reported in 1 participant.
- Cohort 1 and 2: Placebo: Participants received placebo matched tablet orally once daily . Participants in Cohort 1 received placebo for 14 days and participants in Cohort 2 received placebo for 2 days before the study was terminated for safety reasons.
Period: Overall Study
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Started | 7 | 3 | 11 | 9
Completed | 6 | 2 | 0 | 6
Not Completed | 1 | 1 | 11 | 3
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 10 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo | Total
Number analyzed (Participants) | 7 | 3 | 11 | 9 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (8.1) | 50.7 (9.7) | 43.4 (9.8) | 46.8 (9.3) | 46.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 3 | 11 | 9 | 30

OUTCOME MEASURES:

1. Primary Outcome: Baseline of Serum Uric Acid
Description: An elevation in serum uric acid, hyperuricemia, is a prerequisite for the development of gout.
Time Frame: Baseline (pre-dose Day 1)
Population: The full analysis population included all participants randomized and who received at least 1 dose of randomization treatment.
Measure: Mean (Standard Deviation); unit: milligram per deciliter(mg/dL)
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
milligram per deciliter(mg/dL) | 8.800 (1.1402) | 9.100 (0.8185) | 8.991 (0.6549) | 9.278 (0.9536)

2. Primary Outcome: Percent Change From Baseline in Serum Uric Acid Level at 24 Hours Post Dose on Day 14
Time Frame: Day 14 Hour 24
Population: The full analysis population included all participants randomized and who received at least 1 dose of randomization treatment. Number of participants analyzed is number of evaluable participants for this outcome measure. No data due to "Cohort 2: PF-06743649 5 mg" termination after 2 days of dosing.
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 6 | 2 | 0 | 6
percent (%) | -52.891 (6.1661) | -67.480 (1.1498) |  | -1.381 (9.1430)
Statistical Analysis 1: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Test type: Superiority or Other; Bayesian ANCOVA; Mean Difference (Final Values) = -52.550, 90% CI 2-sided [-56.320 to -48.780]
Statistical Analysis 2: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Test type: Superiority or Other; Bayesian ANCOVA; Mean Difference (Final Values) = -66.310, 90% CI 2-sided [-71.310 to -61.540]

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state AEs included both serious and non-serious events.
Time Frame: Baseline up to 28 days after last study drug administration (Day 42)
Population: The safety analysis population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
participants
  Participants with AEs | 2 | 3 | 3 | 4
  Participants with SAEs | 0 | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality. Laboratory test parameters include hematology (Hemoglobin, Hematocrit, red blood cell [RBC] count, Platelet count, mean corpuscular volume [MCV], mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration [MCHC], white blood cell [WBC] count, Total neutrophils, Eosinophils, Monocytes, Basophils, Lymphocytes), hematocrit (blood urea nitrogen [BUN]/urea and Creatinine, Glucose , Calcium, Sodium, Potassium, Chloride, Total CO2 [Bicarbonate], aspartate transaminase [AST], alanine transaminase [ALT], Total Bilirubin, Alkaline phosphatase, Albumin, Total protein, Thyroid Stimulating Hormone [TSH], free T3 [FT3] and free T4 [FT4] ), urinalysis (pH, Glucose [qual], Protein, Blood, Ketones, Nitrites, Leukocyte esterase, Urobilinogen, Urine bilirubin, Microscopy [including crystals]) and other (follicle-stimulating hormone [FSH], Urine drug screen).
Time Frame: Baseline up to follow up visit (Day 25-29)
Population: The safety analysis population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
participants | 1 | 1 | 3 | 2

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Criteria for potential clinically important change in vital signs included: Systolic blood pressure (BP) less than (<) 90 millimeters of mercury (mmHg) or more than or equal to (>=)30 mmHg change from baseline, diastolic BP of <50 mmHg or >=20 mmHg change from baseline, Supine pulse rate of <40 or more than (>)120 beats per minute (bpm).
Time Frame: Baseline up to follow up visit (Day 25-29)
Population: The safety analysis population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
participants
  Supine Systolic BP (mmHg) <90 | 0 | 0 | 0 | 0
  Supine Diastolic BP (mmHg) <50 | 0 | 0 | 0 | 0
  Supine Pulse Rate (bpm) <40 | 0 | 0 | 0 | 0
  Supine Pulse Rate (bpm) >120 | 0 | 0 | 0 | 0
  Increase Supine Systolic BP (mmHg) >=30 | 1 | 0 | 1 | 1
  Increase Supine Diastolic BP (mmHg) >=20 | 1 | 0 | 1 | 1
  Decrease Supine Systolic BP (mmHg) >=30 | 0 | 0 | 1 | 0
  Decrease Supine Diastolic BP (mmHg) >=20 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Values Meeting Categorical Summarization Criteria
Description: Criteria for potential clinically important changes in ECG (12-lead) were defined as: the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization (PR interval) >=300 milliseconds (msec) or increase from baseline >=25% when baseline >200 msec or increase from baseline >=50% when baseline less than or equal to (<=) 200 msec; time from the beginning of the electrocardiogram Q wave to the end of the S wave corresponding to ventricular depolarization (QRS) interval >=140 msec or >=50% increase from baseline; the beginning of the Q wave to the end of the T wave corresponding to electrical systole (QT) interval corrected using the Fridericia formula (QTcF) of 450 to < 480 msec, 480 to <500 msec and >=500 msec, or an increase of 30 to <60 msec or >=60 msec from baseline.
Time Frame: Baseline up to Day 16
Population: The safety analysis population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
participants
  PR (msec) >=300 | 0 | 0 | 0 | 0
  QRS complex (msec) >=140 | 0 | 0 | 0 | 0
  QTCF (msec) 450-<480 | 0 | 0 | 0 | 0
  QTCF (msec) 480-<500 | 0 | 0 | 0 | 0
  QTCF (msec) >=500 | 0 | 0 | 0 | 0
  PR increase from baseline >=25/50% | 0 | 0 | 0 | 0
  QRS complex increase from baseline >=50% | 0 | 0 | 0 | 0
  QTCF increase from baseline 30 to <60 msec | 0 | 0 | 0 | 0
  QTCF increase from baseline >=60 msec | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Serum Uric Acid Levels at Day 1, Day 3, Day 7, Day 11, Day 14 and Follow-up
Time Frame: Day 1, Day 3, Day 7, Day 11, Day 14 and follow-up visit (Day 25-29)
Population: The full analysis population included all participants randomized and who received at least 1 dose of randomization treatment; n=number of participants analyzed in each respective arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
mg/dL
  Baseline (n=7,3,11,9) | 8.80 (1.140) | 9.10 (0.819) | 8.99 (0.655) | 9.28 (0.954)
  Day 1, Hour 1 (n=6,3,11, 9) | -0.18 (0.194) | -0.50 (0.436) | -0.51 (0.353) | 0.11 (0.190)
  Day 1, Hour 2 (n=7,3,11,9) | -0.69 (0.261) | -1.17 (0.839) | -1.27 (0.403) | -0.02 (0.156)
  Day 1, Hour 4 (n=7,3,11,9) | -1.47 (0.293) | -3.07 (0.115) | -2.30 (0.382) | -0.12 (0.233)
  Day 1, Hour 8 (n=7,3,11,9) | -2.00 (0.716) | -3.87 (0.473) | -2.77 (0.623) | -0.23 (0.320)
  Day 1, Hour 12 (n=7,3,11,9) | -1.77 (0.704) | -3.83 (0.577) | -2.74 (0.721) | -0.19 (0.389)
  Day 1, Hour 24 (n=7,3,11,9) | -1.69 (0.664) | -3.43 (0.757) | -2.04 (0.770) | -0.18 (0.396)
  Day 3 (n=7,3,10,9) | -2.13 (0.921) | -4.50 (0.529) | -3.02 (0.925) | 0.08 (0.342)
  Day 7, pre-dose (n=7,2,0,6) | -2.60 (0.945) | -5.75 (0.212) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.07 (0.734)
  Day 7, Hour 1 (n=7,2,0,6) | -2.64 (0.846) | -5.75 (0.212) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.03 (0.787)
  Day 7, Hour 2 (n=7,2,0,6) | -2.94 (0.838) | -6.10 (0.283) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.05 (0.797)
  Day 7, Hour 4 (n=7,2,0,6) | -3.44 (0.873) | -6.60 (0.283) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.22 (0.731)
  Day 7, Hour 8 (n=7,2,0,6) | -3.49 (0.996) | -6.60 (0.141) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.38 (0.578)
  Day 7, Hour 12 (n=7,2,0,6) | -3.24 (1.037) | -6.45 (0.071) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.25 (0.599)
  Day 7, Hour 24 (n=7,2,0,6) | -2.73 (0.955) | -5.90 (0.141) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.17 (0.794)
  Day 11 (n=6,2,0,6) | -4.80 (0.961) | -5.75 (0.071) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.17 (0.845)
  Day 14, pre-dose (n=6,2,0,6) | -4.57 (0.900) | -5.75 (0.636) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.22 (0.747)
  Day 14, Hour 1 (n=6,2,0,6) | -4.83 (0.799) | -6.05 (0.495) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.23 (0.659)
  Day 14, Hour 2 (n=6,2,0,6) | -5.35 (0.846) | -6.35 (0.495) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.33 (0.680)
  Day 14, Hour 4 (n=6,2,0,6) | -6.02 (0.906) | -6.80 (0.566) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.55 (0.638)
  Day 14, Hour 8 (n=6,2,0,6) | -5.93 (1.001) | -6.85 (0.636) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.33 (0.781)
  Day 14, Hour 12 (n=6,2,0,6) | -5.67 (1.124) | -6.60 (0.566) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.28 (0.725)
  Day 14, Hour 24 (n=6,2,0,6) | -4.85 (0.940) | -5.90 (0.424) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.20 (0.834)
  Follow-up (Day 25-29) (n=6,3,10,9) | -0.93 (1.422) | -2.27 (2.593) | 0.45 (0.938) | -0.30 (1.648)
Statistical Analysis 1: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.30, 90% CI [-0.55 to -0.06], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.62, 90% CI 2-sided [-0.95 to -0.28], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -1.34, 90% CI 2-sided [-1.52 to -1.16], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -1.86, 90% CI 2-sided [-2.38 to -1.33], Standard Error of Mean 0.29
Statistical Analysis 5: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -1.83, 90% CI 2-sided [-2.18 to -1.48], Standard Error of Mean 0.19
Statistical Analysis 6: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -1.74, 90% CI 2-sided [-2.11 to -1.37], Standard Error of Mean 0.20
Statistical Analysis 7: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 3; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -2.48, 90% CI 2-sided [-2.89 to -2.06], Standard Error of Mean 0.23
Statistical Analysis 8: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -2.75, 90% CI 2-sided [-3.29 to -2.20], Standard Error of Mean 0.30
Statistical Analysis 9: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -2.80, 90% CI 2-sided [-3.39 to -2.21], Standard Error of Mean 0.33
Statistical Analysis 10: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -3.06, 90% CI 2-sided [-3.72 to -2.41], Standard Error of Mean 0.36
Statistical Analysis 11: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day7, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -3.40, 90% CI 2-sided [-4.03 to -2.77], Standard Error of Mean 0.35
Statistical Analysis 12: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -3.30, 90% CI 2-sided [-3.82 to -2.79], Standard Error of Mean 0.28
Statistical Analysis 13: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -3.20, 90% CI 2-sided [-3.72 to -2.68], Standard Error of Mean 0.28
Statistical Analysis 14: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -2.81, 90% CI 2-sided [-3.30 to -2.32], Standard Error of Mean 0.27
Statistical Analysis 15: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 11; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -4.56, 90% CI 2-sided [-5.19 to -3.92], Standard Error of Mean 0.35
Statistical Analysis 16: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -4.32, 90% CI 2-sided [-4.75 to -3.88], Standard Error of Mean 0.23
Statistical Analysis 17: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -4.55, 90% CI 2-sided [-5.02 to -4.08], Standard Error of Mean 0.25
Statistical Analysis 18: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -4.97, 90% CI 2-sided [-5.47 to -4.47], Standard Error of Mean 0.27
Statistical Analysis 19: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -5.43, 90% CI 2-sided [-5.83 to -5.02], Standard Error of Mean 0.22
Statistical Analysis 20: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -5.57, 90% CI 2-sided [-6.08 to -5.05], Standard Error of Mean 0.28
Statistical Analysis 21: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -5.34, 90% CI 2-sided [-5.86 to -4.82], Standard Error of Mean 0.28
Statistical Analysis 22: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -4.65, 90% CI 2-sided [-5.12 to -4.18], Standard Error of Mean 0.25
Statistical Analysis 23: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Follow-up, Day 25-29; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -1.09, 90% CI 2-sided [-2.97 to 0.79], Standard Error of Mean 1.03
Statistical Analysis 24: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.62, 90% CI 2-sided [-0.92 to -0.32], Standard Error of Mean 0.17
Statistical Analysis 25: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -1.18, 90% CI 2-sided [-1.61 to -0.75], Standard Error of Mean 0.24
Statistical Analysis 26: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -2.91, 90% CI 2-sided [-3.14 to -2.69], Standard Error of Mean 0.12
Statistical Analysis 27: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -3.70, 90% CI 2-sided [-4.36 to -3.03], Standard Error of Mean 0.37
Statistical Analysis 28: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -3.84, 90% CI 2-sided [-4.28 to -3.40], Standard Error of Mean 0.24
Statistical Analysis 29: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -3.47, 90% CI [-3.94 to -3.00], Standard Error of Mean 0.26
Statistical Analysis 30: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 3; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -4.76, 90% CI 2-sided [-5.29 to -4.23], Standard Error of Mean 0.29
Statistical Analysis 31: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -5.81, 90% CI 2-sided [-6.62 to -5.00], Standard Error of Mean 0.45
Statistical Analysis 32: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -5.84, 90% CI 2-sided [-6.72 to -4.95], Standard Error of Mean 0.49
Statistical Analysis 33: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -6.18, 90% CI 2-sided [-7.17 to -5.19], Standard Error of Mean 0.55
Statistical Analysis 34: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -6.51, 90% CI 2-sided [-7.46 to -5.55], Standard Error of Mean 0.53
Statistical Analysis 35: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -6.29, 90% CI 2-sided [-7.07 to -5.51], Standard Error of Mean 0.43
Statistical Analysis 36: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -6.24, 90% CI 2-sided [-7.03 to -5.44], Standard Error of Mean 0.44
Statistical Analysis 37: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -5.75, 90% CI 2-sided [-6.50 to -4.99], Standard Error of Mean 0.42
Statistical Analysis 38: Comparison: Cohort 1: PF-06743649 40 mg; Day 11; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -5.62, 90% CI 2-sided [-6.59 to -4.65], Standard Error of Mean 0.53
Statistical Analysis 39: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -5.76, 90% CI 2-sided [-6.42 to -5.10], Standard Error of Mean 0.36
Statistical Analysis 40: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -5.96, 90% CI 2-sided [-6.67 to -5.24], Standard Error of Mean 0.39
Statistical Analysis 41: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -6.14, 90% CI 2-sided [-6.90 to -5.38], Standard Error of Mean 0.41
Statistical Analysis 42: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -6.42, 90% CI 2-sided [-7.03 to -5.81], Standard Error of Mean 0.33
Statistical Analysis 43: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -6.64, 90% CI 2-sided [-7.41 to -5.87], Standard Error of Mean 0.42
Statistical Analysis 44: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -6.40, 90% CI 2-sided [-7.18 to -5.63], Standard Error of Mean 0.42
Statistical Analysis 45: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -5.77, 90% CI 2-sided [-6.47 to -5.07], Standard Error of Mean 0.38
Statistical Analysis 46: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Follow-up, Day 25-29; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -2.66, 90% CI 2-sided [-4.96 to -0.35], Standard Error of Mean 1.26

8. Secondary Outcome: Number of Participants Reaching Serum Uric Acid Levels <6, <5 and <4 mg/dL at 24 Hours Post Dose on Day 7 and Day 14
Description: Number of participants reaching serum uric acid levels <6, <5 and <4 mg/dL at 7 and 14 days after initiation.
Time Frame: 24 hours post dose on Day 7 and Day 14
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 0 | 9
participants
  Day 7 (<6.0) | 4 | 2 |  | 0
  Day 7 (<5.0) | 0 | 2 |  | 0
  Day 7 (<4.0) | 0 | 2 |  | 0
  Day 14 (<6.0) | 6 | 2 |  | 0
  Day 14 (<5.0) | 6 | 2 |  | 0
  Day 14 (<4.0) | 1 | 2 |  | 0

9. Secondary Outcome: Incidence and Severity of Gout Flare Attacks
Time Frame: Baseline up to Day 42
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Duration of Gout Flare Attacks
Description: Duration of gout flare attacks with participants who developed gout flare attacks.
Time Frame: Baseline up to Day 42
Population: Participants who developed gout flare attacks (Duration was not assessed as no participant developed gout flare attacks).
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Plasma Levels of PF-06743649 After Initiation of Dosing at Day 1, Day 7, and Day 14
Description: Data has been calculated by setting concentration values below the lower limit of quantification to zero. The lower limit of quantification was 10.0 nanograms per milliliter (ng/mL).
Time Frame: 0, 1, 2, 4, 8, 12 and 24 hours at Day 1, Day 7, and Day 14
Population: All participants randomized and treated who have at least 1 measureable concentration; n=number of participants analyzed in each respective arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg
Number analyzed (Participants) | 7 | 3 | 11
ng/mL
  Day 1, Hour 0 (n=7,3,11) | NA (NA) — Data was not reported because the observations were not above lower limit of quantification. | NA (NA) — Data was not reported because the observations were not above lower limit of quantification. | NA (NA) — Data was not reported because the observations were not above lower limit of quantification.
  Day 1, Hour 1 (n=7,3,11) | 163.8 (84.336) | 1097 (1011.8) | 371.3 (239.52)
  Day 1, Hour 2 (n=7,3,11) | 196.6 (47.367) | 1570 (416.77) | 454.7 (141.62)
  Day 1, Hour 4 (n=7,3,11) | 105.8 (34.342) | 1081 (189.22) | 282.4 (106.48)
  Day 1, Hour 8 (n=7,3,11) | 47.27 (19.596) | 523.3 (108.89) | 142.7 (87.111)
  Day 1, Hour 12 (n=7,3,11) | 26.84 (13.738) | 229.3 (36.665) | 99.27 (70.301)
  Day 1, Hour 24 (n=7,3,11) | 7.586 (10.183) | 86.67 (18.434) | 48.90 (49.583)
  Day 7, Hour 0 (n=7,2,0) | 10.50 (10.560) | 154.0 (41.012) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 1 (n=7,2,0) | 185.9 (102.26) | 1275 (261.63) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 2 (n=7,2,0) | 211.7 (95.552) | 2715 (487.90) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 4 (n=7,2,0) | 137.3 (43.222) | 1520 (183.85) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 8 (n=7,2,0) | 67.59 (19.509) | 697.0 (49.497) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 12 (n=7,2,0) | 42.30 (16.272) | 457.5 (78.489) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 24 (n=7,2,0) | 12.50 (10.356) | 147.0 (31.113) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 0 (n=6,2,0) | 47.08 (27.363) | 157.5 (43.134) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 1 (n=6,2,0) | 736.7 (483.18) | 1995 (417.19) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 2 (n=6,2,0) | 729.5 (218.79) | 2140 (325.27) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 4 (n=6,2,0) | 429.5 (165.51) | 1480 (325.27) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 8 (n=6,2,0) | 245.8 (99.385) | 687.0 (96.167) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 12 (n=6,2,0) | 163.3 (73.480) | 400.0 (74.953) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 24 (n=6,2,0) | 54.27 (34.849) | 133.5 (13.435) | NA (NA) — No data due to cohort termination after 2 days of dosing.

12. Secondary Outcome: Plasma Levels of PF-06743648 After Initiation of Dosing at Day 1, Day 7, and Day 14
Description: PF-06743648 is an active metabolite of PF-06743649. Data has been calculated by setting concentration values below the lower limit of quantification to zero. The lower limit of quantification was 2.00 nanograms per milliliter (ng/mL).
Time Frame: Day 1, Day 7, and Day 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg
Number analyzed (Participants) | 7 | 3 | 11
ng/mL
  Day 1, Hour 0 (n=7,3,11) | NA (NA) — Data was not reported because the observations were not above lower limit of quantification. | NA (NA) — Data was not reported because the observations were not above lower limit of quantification. | NA (NA) — Data was not reported because the observations were not above lower limit of quantification.
  Day 1, Hour 1 (n=7,3,11) | 6.713 (6.6738) | 79.62 (82.093) | 13.81 (10.519)
  Day 1, Hour 2 (n=7,3,11) | 28.69 (14.265) | 245.6 (182.75) | 49.30 (26.599)
  Day 1, Hour 4 (n=7,3,11) | 30.07 (7.3081) | 395.0 (69.936) | 59.21 (29.231)
  Day 1, Hour 8 (n=7,3,11) | 18.09 (5.4462) | 261.3 (53.003) | 38.25 (18.527)
  Day 1, Hour 12 (n=7,3,11) | 11.46 (3.4996) | 156.3 (22.591) | 25.67 (13.251)
  Day 1, Hour 24 (n=7,3,11) | 6.059 (2.8621) | 76.27 (23.811) | 12.76 (7.3997)
  Day 7, Hour 0 (n=7,2,0) | 7.259 (3.5055) | 70.50 (11.597) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 1 (n=7,2,0) | 22.00 (9.8895) | 107.0 (1.4142) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 2 (n=7,2,0) | 42.83 (20.763) | 344.0 (49.497) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 4 (n=7,2,0) | 40.26 (13.353) | 397.0 (9.8995) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 8 (n=7,2,0) | 26.64 (9.2428) | 261.0 (0.00000) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 12 (n=7,2,0) | 16.67 (5.5011) | 167.5 (23.335) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 7, Hour 24 (n=7,2,0) | 8.470 (3.7998) | 91.80 (1.9799) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 0 (n=6,2,0) | 21.99 (9.6890) | 76.60 (9.4752) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 1 (n=6,2,0) | 74.72 (37.910) | 171.0 (26.870) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 2 (n=6,2,0) | 139.3 (53.432) | 390.0 (117.38) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 4 (n=6,2,0) | 127.3 (37.255) | 364.0 (18.385) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 8 (n=6,2,0) | 74.82 (39.810) | 280.5 (9.1924) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 12 (n=6,2,0) | 49.07 (27.960) | 162.0 (1.4142) | NA (NA) — No data due to cohort termination after 2 days of dosing.
  Day 14, Hour 24 (n=6,2,0) | 27.32 (14.608) | 81.35 (1.2021) | NA (NA) — No data due to cohort termination after 2 days of dosing.

13. Secondary Outcome: Change From Baseline in Plasma Levels of Xanthine at Day 1, Day 7, Day 14, and at Follow-up
Description: Change in plasma levels of xanthine from baseline at time points 0 (prior to dosing except on Day 1), 1, 2, 4, 8, 12 and 24 hours following dosing with PF-06743649 or placebo on days 1, 7 and 14 as well prior to dosing on days 3 and 11 and at follow-up of treatment with PF-06743649 or placebo.
Time Frame: Baseline, Day 1, Day 7, Day 14, and at follow-up visit (Day 25-29)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
micrograms per milliliter (mcg/mL)
  Baseline (n=7,3,11,9) | 0.2519 (0.04316) | 0.2680 (0.10095) | 0.2102 (0.04037) | 0.2257 (0.05304)
  Day 1, Hour 1 (n=7,3,11,9) | -0.0473 (0.05949) | 0.1057 (0.02155) | -0.0192 (0.04214) | -0.0112 (0.08230)
  Day 1, Hour 2 (n=7,3,11,9) | -0.0330 (0.03844) | 0.3667 (0.27216) | 0.0346 (0.05090) | -0.0220 (0.03653)
  Day 1, Hour 4 (n=7,3,11,9) | -0.0826 (0.04922) | 0.3317 (0.11558) | -0.0306 (0.05783) | -0.0511 (0.06510)
  Day 1, Hour 8 (n=7,3,11,9) | -0.0859 (0.07603) | 0.1947 (0.14431) | -0.0918 (0.02295) | -0.0982 (0.3674)
  Day 1, Hour 12 (n=7,3,11,9) | -0.1117 (0.04270) | 0.0847 (0.11634) | -0.0921 (0.03801) | -0.0786 (0.05731)
  Day 1, Hour 24 (n=7,3,11,9) | 0.0167 (0.08149) | 0.1927 (0.04879) | 0.0140 (0.03411) | 0.0233 (0.10687)
  Day 7, pre-dose (n=7,2,0,6) | -0.0362 (0.07118) | 0.1450 (0.00283) | NA (NA) — No data due to cohort termination after 2 days of dosing. | 0.0177 (0.13598)
  Day 7, Hour 1 (n=7,2,0,6) | -0.0061 (0.10488) | 0.1765 (0.07566) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0170 (0.07475)
  Day 7, Hour 2 (n=7,2,0,6) | 0.0231 (0.05070) | 0.5300 (0.21779) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0098 (0.08066)
  Day 7, Hour 4 (n=7,2,0,6) | -0.0147 (0.06839) | 0.4995 (0.14920) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0233 (0.07942)
  Day 7, Hour 8 (n=7,2,0,6) | -0.1086 (0.04749) | 0.3010 (0.14425) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0843 (0.05064)
  Day 7, Hour 12 (n=7,2,0,6) | -0.1276 (0.04658) | -0.0535 (0.01909) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0750 (0.04685)
  Day 7, Hour 24 (n=7,2,0,6) | -0.0540 (0.05434) | 0.1465 (0.07990) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0242 (0.06072)
  Day 14, pre-dose (n=6,2,0,6) | -0.0290 (0.05418) | 0.1540 (0.07778) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0120 (0.02367)
  Day 14, Hour 1 (n=6,2,0,6) | 0.0607 (0.06662) | 0.3515 (0.10819) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0008 (0.02699)
  Day 14, Hour 2 (n=6,2,0,6) | 0.1353 (0.09010) | 0.5960 (0.01131) | NA (NA) — No data due to cohort termination after 2 days of dosing. | 0.0330 (0.09579)
  Day 14, Hour 4 (n=6,2,0,6) | -0.0148 (0.09997) | 0.5595 (0.00212) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0210 (0.07869)
  Day 14, Hour 8 (n=6,2,0,6) | -0.0655 (0.08041) | 0.2030 (0.11738) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0778 (0.06107)
  Day 14, Hour 12 (n=6,2,0,6) | -0.0986 (0.04973) | 0.1175 (0.18031) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0801 (0.04477)
  Day 14, Hour 24 (n=6,2,0,6) | -0.0172 (0.08536) | 0.1695 (0.08132) | NA (NA) — No data due to cohort termination after 2 days of dosing. | 0.0242 (0.06158)
  Follow-up (Day 25-29) (n=6,3,10,9) | 0.3710 (0.92324) | 0.8263 (0.77448) | 0.1161 (0.18229) | 0.2299 (0.44888)
Statistical Analysis 1: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0355, 90% CI 2-sided [-0.1103 to 0.0394], Standard Error of Mean 0.0423
Statistical Analysis 2: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0152, 90% CI 2-sided [-0.1269 to 0.0966], Standard Error of Mean 0.0631
Statistical Analysis 3: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0331, 90% CI 2-sided [-0.1078 to 0.0417], Standard Error of Mean 0.0422
Statistical Analysis 4: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.0035, 90% CI 2-sided [-0.0750 to 0.0820], Standard Error of Mean 0.0443
Statistical Analysis 5: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0502, 90% CI 2-sided [-0.1153 to 0.0149], Standard Error of Mean 0.0367
Statistical Analysis 6: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0080, 90% CI 2-sided [-0.1058 to 0.0899], Standard Error of Mean 0.0553
Statistical Analysis 7: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0539, 90% CI 2-sided [-0.1538 to 0.0460], Standard Error of Mean 0.0561
Statistical Analysis 8: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.0109, 90% CI 2-sided [-0.0793 to 0.1010], Standard Error of Mean 0.0506
Statistical Analysis 9: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.0330, 90% CI 2-sided [-0.0554 to 0.1213], Standard Error of Mean 0.0496
Statistical Analysis 10: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.0086, 90% CI 2-sided [-0.0733 to 0.0905], Standard Error of Mean 0.0459
Statistical Analysis 11: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0244, 90% CI 2-sided [-0.0865 to 0.0378], Standard Error of Mean 0.0349
Statistical Analysis 12: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0526, 90% CI 2-sided [-0.0973 to -0.0079], Standard Error of Mean 0.0251
Statistical Analysis 13: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0298, 90% CI 2-sided [-0.0889 to 0.0292], Standard Error of Mean 0.0331
Statistical Analysis 14: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0167, 90% CI 2-sided [-0.0649 to 0.0315], Standard Error of Mean 0.0268
Statistical Analysis 15: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.0616, 90% CI 2-sided [0.0010 to 0.1222], Standard Error of Mean 0.0337
Statistical Analysis 16: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.1025, 90% CI 2-sided [0.0104 to 0.1945], Standard Error of Mean 0.0512
Statistical Analysis 17: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.0062, 90% CI 2-sided [-0.0827 to 0.0952], Standard Error of Mean 0.0495
Statistical Analysis 18: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.0124, 90% CI 2-sided [-0.0672 to 0.0919], Standard Error of Mean 0.0443
Statistical Analysis 19: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0186, 90% CI 2-sided [-0.0918 to 0.0547], Standard Error of Mean 0.0408
Statistical Analysis 20: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.0413, 90% CI 2-sided [-0.1192 to 0.0365], Standard Error of Mean 0.0433
Statistical Analysis 21: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Follow-up, Day 25-29; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.4011, 90% CI 2-sided [-0.2968 to 1.0990], Standard Error of Mean 0.3916
Statistical Analysis 22: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.1175, 90% CI 2-sided [0.0223 to 0.2127], Standard Error of Mean 0.0537
Statistical Analysis 23: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.3845, 90% CI 2-sided [0.2424 to 0.5266], Standard Error of Mean 0.0802
Statistical Analysis 24: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.3812, 90% CI 2-sided [0.2862 to 0.4762], Standard Error of Mean 0.0536
Statistical Analysis 25: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.2841, 90% CI 2-sided [0.1843 to 0.3838], Standard Error of Mean 0.0563
Statistical Analysis 26: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.1462, 90% CI 2-sided [0.0635 to 0.2289], Standard Error of Mean 0.0467
Statistical Analysis 27: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.1680, 90% CI 2-sided [0.0436 to 0.2924], Standard Error of Mean 0.0702
Statistical Analysis 28: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.1303, 90% CI 2-sided [-0.0172 to 0.2778], Standard Error of Mean 0.0830
Statistical Analysis 29: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.1953, 90% CI [0.0625 to 0.3281], Standard Error of Mean 0.0747
Statistical Analysis 30: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.5409, 90% CI 2-sided [0.4110 to 0.6707], Standard Error of Mean 0.0729
Statistical Analysis 31: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.5235, 90% CI 2-sided [0.4032 to 0.6438], Standard Error of Mean 0.0675
Statistical Analysis 32: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.3857, 90% CI 2-sided [0.2944 to 0.4769], Standard Error of Mean 0.0512
Statistical Analysis 33: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.0216, 90% CI 2-sided [-0.0439 to 0.0872], Standard Error of Mean 0.0368
Statistical Analysis 34: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.1708, 90% CI 2-sided [0.0841 to 0.2574], Standard Error of Mean 0.0486
Statistical Analysis 35: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.1660, 90% CI 2-sided [0.0982 to 0.2338], Standard Error of Mean 0.0377
Statistical Analysis 36: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.3524, 90% CI 2-sided [0.2667 to 0.4380], Standard Error of Mean 0.0477
Statistical Analysis 37: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.5631, 90% CI 2-sided [0.4330 to 0.6932], Standard Error of Mean 0.0724
Statistical Analysis 38: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.5807, 90% CI 2-sided [0.4549 to 0.7065], Standard Error of Mean 0.0700
Statistical Analysis 39: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.2814, 90% CI 2-sided [0.1688 to 0.3940], Standard Error of Mean 0.0627
Statistical Analysis 40: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.1982, 90% CI 2-sided [0.0945 to 0.3019], Standard Error of Mean 0.0577
Statistical Analysis 41: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.1465, 90% CI 2-sided [0.0361 to 0.2569], Standard Error of Mean 0.0615
Statistical Analysis 42: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Follow-up, Day 25-29; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.8565, 90% CI 2-sided [0.0017 to 1.7112], Standard Error of Mean 0.4796

14. Secondary Outcome: Change From Baseline in Plasma Levels of Hypoxanthine at Day 1, Day 7, Day 14, and at Follow-up
Time Frame: Day 1, Day 7, Day 14, and at follow-up visit (Day 25-29)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
mcg/mL
  Baseline (n=7,3,11,9) | 0.9604 (0.15380) | 1.0060 (0.41079) | 0.8677 (0.18896) | 0.8922 (0.13486)
  Day 1, Hour 1 (n=7,3,11,9) | -0.2539 (0.24173) | 0.1440 (0.56564) | -0.1205 (0.16427) | 0.0847 (0.41097)
  Day 1, Hour 2 (n=7,3,11,9) | -0.2229 (0.08132) | 0.2130 (0.40812) | -0.0145 (0.13714) | -0.0421 (0.21113)
  Day 1, Hour 4 (n=7,3,11,9) | -0.2774 (0.19696) | 0.0717 (0.62608) | -0.1426 (0.14932) | -0.0369 (0.32185)
  Day 1, Hour 8 (n=7,3,11,9) | -0.2000 (0.27433) | 0.1760 (0.78402) | -0.1895 (0.18641) | -0.1870 (0.26137)
  Day 1, Hour 12 (n=7,3,11,9) | -0.2973 (0.13666) | 0.2703 (0.62935) | -0.0979 (0.15883) | -0.0967 (0.22579)
  Day 1, Hour 24 (n=7,3,11,9) | -0.0937 (0.30529) | 0.5607 (0.66507) | -0.0039 (0.10751) | 0.1200 (0.48900)
  Day 7, pre-dose (n=7,2,0,6) | -0.1309 (0.31653) | 0.0810 (0.21355) | NA (NA) — No data due to cohort termination after 2 days of dosing. | 0.1317 (0.57974)
  Day 7, Hour 1 (n=7,2,0,6) | -0.1089 (0.40558) | -0.1575 (0.46598) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0285 (0.43096)
  Day 7, Hour 2 (n=7,2,0,6) | -0.0923 (0.11659) | 0.1360 (0.67317) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0103 (0.35162)
  Day 7, Hour 4 (n=7,2,0,6) | -0.0067 (0.28262) | -0.2505 (0.37406) | NA (NA) — No data due to cohort termination after 2 days of dosing. | 0.0762 (0.37371)
  Day 7, Hour 8 (n=7,2,0,6) | -0.2610 (0.30443) | -0.0495 (0.61023) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0543 (0.35172)
  Day 7, Hour 12 (n=7,2,0,6) | -0.2860 (0.21522) | -0.5290 (0.32951) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.1557 (0.15279)
  Day 7, Hour 24 (n=7,2,0,6) | -0.1926 (0.18082) | 0.1410 (0.68024) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0680 (0.35421)
  Day 14, pre-dose (n=6,2,0,6) | -0.2573 (0.23823) | 0.0710 (0.24183) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0978 (0.10319)
  Day 14, Hour 1 (n=6,2,0,6) | -0.2292 (0.13816) | 0.1660 (0.30547) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.1065 (0.19276)
  Day 14, Hour 2 (n=6,2,0,6) | -0.1970 (0.20110) | 0.2860 (0.29133) | NA (NA) — No data due to cohort termination after 2 days of dosing. | 0.0047 (0.25228)
  Day 14, Hour 4 (n=6,2,0,6) | -0.3627 (0.22065) | 0.1210 (0.42568) | NA (NA) — No data due to cohort termination after 2 days of dosing. | 0.0133 (0.30407)
  Day 14, Hour 8 (n=6,2,0,6) | -0.2898 (0.32120) | -0.2310 (0.16829) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.0698 (0.34513)
  Day 14, Hour 12 (n=6,2,0,6) | -0.2415 (0.19015) | 0.0510 (0.11455) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.1075 (0.20019)
  Day 14, Hour 24 (n=6,2,0,6) | -0.2030 (0.23638) | 0.2260 (0.36204) | NA (NA) — No data due to cohort termination after 2 days of dosing. | 0.0855 (0.36310)
  Follow-up Day 25-29 (n=6,3,10,9) | -0.0965 (0.43007) | -0.2550 (0.91149) | 0.3204 (0.30373) | 0.3778 (0.73741)
Statistical Analysis 1: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.348, 90% CI 2-sided [-0.707 to 0.010], Standard Error of Mean 0.209
Statistical Analysis 2: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.179, 90% CI 2-sided [-0.533 to 0.175], Standard Error of Mean 0.205
Statistical Analysis 3: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.258, 90% CI 2-sided [-0.568 to 0.052], Standard Error of Mean 0.180
Statistical Analysis 4: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.046, 90% CI [-0.390 to 0.298], Standard Error of Mean 0.201
Statistical Analysis 5: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.284, 90% CI [-0.575 to 0.006], Standard Error of Mean 0.168
Statistical Analysis 6: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.166, 90% CI 2-sided [-0.569 to 0.237], Standard Error of Mean 0.235
Statistical Analysis 7: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.263, 90% CI 2-sided [-0.657 to 0.132], Standard Error of Mean 0.230
Statistical Analysis 8: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.080, 90% CI 2-sided [-0.460 to 0.299], Standard Error of Mean 0.221
Statistical Analysis 9: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.082, 90% CI 2-sided [-0.392 to 0.228], Standard Error of Mean 0.180
Statistical Analysis 10: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.083, 90% CI 2-sided [-0.408 to 0.242], Standard Error of Mean 0.189
Statistical Analysis 11: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.207, 90% CI 2-sided [-0.508 to 0.095], Standard Error of Mean 0.174
Statistical Analysis 12: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.130, 90% CI 2-sided [-0.451 to 0.191], Standard Error of Mean 0.186
Statistical Analysis 13: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.125, 90% CI 2-sided [-0.445 to 0.196], Standard Error of Mean 0.186
Statistical Analysis 14: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.188, 90% CI 2-sided [-0.472 to 0.097], Standard Error of Mean 0.162
Statistical Analysis 15: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.152, 90% CI 2-sided [-0.434 to 0.130], Standard Error of Mean 0.161
Statistical Analysis 16: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.231, 90% CI 2-sided [-0.504 to 0.043], Standard Error of Mean 0.155
Statistical Analysis 17: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.405, 90% CI 2-sided [-0.722 to -0.088], Standard Error of Mean 0.184
Statistical Analysis 18: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.249, 90% CI 2-sided [-0.560 to 0.062], Standard Error of Mean 0.180
Statistical Analysis 19: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.163, 90% CI 2-sided [-0.467 to 0.141], Standard Error of Mean 0.176
Statistical Analysis 20: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.317, 90% CI 2-sided [-0.633 to -0.002], Standard Error of Mean 0.183
Statistical Analysis 21: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Follow-up, Day 25-29; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.094, 90% CI 2-sided [-0.683 to 0.496], Standard Error of Mean 0.339
Statistical Analysis 22: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.050, 90% CI 2-sided [-0.406 to 0.505], Standard Error of Mean 0.266
Statistical Analysis 23: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.257, 90% CI 2-sided [-0.193 to 0.707], Standard Error of Mean 0.260
Statistical Analysis 24: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.091, 90% CI 2-sided [-0.302 to 0.485], Standard Error of Mean 0.229
Statistical Analysis 25: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.330, 90% CI 2-sided [-0.107 to 0.768], Standard Error of Mean 0.256
Statistical Analysis 26: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.283, 90% CI 2-sided [-0.087 to 0.653], Standard Error of Mean 0.214
Statistical Analysis 27: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.488, 90% CI 2-sided [-0.024 to 1.000], Standard Error of Mean 0.299
Statistical Analysis 28: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.206, 90% CI 2-sided [-0.356 to 0.768], Standard Error of Mean 0.327
Statistical Analysis 29: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.123, 90% CI 2-sided [-0.410 to 0.656], Standard Error of Mean 0.310
Statistical Analysis 30: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.396, 90% CI 2-sided [-0.025 to 0.818], Standard Error of Mean 0.246
Statistical Analysis 31: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.077, 90% CI 2-sided [-0.523 to 0.368], Standard Error of Mean 0.260
Statistical Analysis 32: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.254, 90% CI 2-sided [-0.154 to 0.661], Standard Error of Mean 0.237
Statistical Analysis 33: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.125, 90% CI 2-sided [-0.564 to 0.315], Standard Error of Mean 0.256
Statistical Analysis 34: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.458, 90% CI 2-sided [0.019 to 0.897], Standard Error of Mean 0.256
Statistical Analysis 35: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, pre-dose; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.418, 90% CI 2-sided [0.043 to 0.792], Standard Error of Mean 0.215
Statistical Analysis 36: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.521, 90% CI 2-sided [0.150 to 0.893], Standard Error of Mean 0.213
Statistical Analysis 37: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 2; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.530, 90% CI 2-sided [0.172 to 0.888], Standard Error of Mean 0.204
Statistical Analysis 38: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 4; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.357, 90% CI 2-sided [-0.069 to 0.782], Standard Error of Mean 0.247
Statistical Analysis 39: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 8; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.088, 90% CI 2-sided [-0.328 to 0.503], Standard Error of Mean 0.242
Statistical Analysis 40: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 12; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.406, 90% CI 2-sided [0.000 to 0.812], Standard Error of Mean 0.236
Statistical Analysis 41: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14, Hour 24; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.377, 90% CI 2-sided [-0.047 to 0.802], Standard Error of Mean 0.247
Statistical Analysis 42: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Follow-up, Day 25-29; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -0.223, 90% CI 2-sided [-0.949 to 0.502], Standard Error of Mean 0.418

15. Secondary Outcome: Change From Baseline in Urinary Uric Acid Levels at Day 1, Day 7, and Day 14
Description: Change from baseline in urinary uric acid cumulative amounts.
Time Frame: Baseline, Day 1, Day 7 and Day 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
mg
  Baseline (n=7,3,11,9) | 658.495 (192.7457) | 745.574 (262.1465) | 590.951 (195.9763) | 583.854 (147.2471)
  Change at Day 1 (n=7,3,11,9) | 308.363 (320.3229) | 424.684 (475.6851) | 168.996 (339.0577) | -19.228 (117.2680)
  Change at Day 7 (n=7,2,0,6) | 38.603 (160.1758) | -28.477 (235.2700) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -23.369 (141.1305)
  Change at Day 14 (n=6,2,0,6) | 55.610 (236.5787) | -79.793 (195.2251) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -34.863 (81.4321)
Statistical Analysis 1: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 316.89, 90% CI 2-sided [21.91 to 611.88], Standard Error of Mean 166.57
Statistical Analysis 2: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 61.97, 90% CI 2-sided [-94.87 to 218.82], Standard Error of Mean 88.27
Statistical Analysis 3: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 107.96, 90% CI 2-sided [-71.20 to 287.11], Standard Error of Mean 100.38
Statistical Analysis 4: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 433.21, 90% CI 2-sided [58.30 to 808.13], Standard Error of Mean 211.71
Statistical Analysis 5: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 13.20, 90% CI 2-sided [-208.07 to 234.47], Standard Error of Mean 125.47
Statistical Analysis 6: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = -29.83, 90% CI 2-sided [-285.26 to 225.60], Standard Error of Mean 142.95

16. Secondary Outcome: Change From Baseline in Urinary Xanthine Levels at Day 1, Day 7, and Day 14
Description: Change from baseline in urinary xanthine cumulative amounts.
Time Frame: Baseline, Day 1, Day 7 and Day 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
mg
  Baseline (n=7,3,11,9) | 7.014 (1.9431) | 8.783 (2.2772) | 5.756 (2.3429) | 6.431 (2.4413)
  Change at Day 1 (n=7,3,11,9) | 3.528 (2.6662) | 13.209 (4.8900) | 1.793 (2.2691) | 0.031 (0.8807)
  Change at Day 7 (n=7,2,0,6) | 2.838 (1.8937) | 27.886 (1.1209) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.832 (1.3666)
  Change at Day 14 (n=6,2,0,6) | 7.291 (2.1068) | 29.063 (2.9613) | NA (NA) — No data due to cohort termination after 2 days of dosing. | -0.708 (0.7644)
Statistical Analysis 1: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 3.44, 90% CI 2-sided [0.71 to 6.17], Standard Error of Mean 1.57
Statistical Analysis 2: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 3.67, 90% CI 2-sided [1.97 to 5.37], Standard Error of Mean 0.94
Statistical Analysis 3: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 8.10, 90% CI 2-sided [6.24 to 9.96], Standard Error of Mean 1.03
Statistical Analysis 4: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 13.12, 90% CI 2-sided [9.65 to 16.59], Standard Error of Mean 2.00
Statistical Analysis 5: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 27.99, 90% CI 2-sided [25.49 to 30.49], Standard Error of Mean 1.40
Statistical Analysis 6: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 28.77, 90% CI 2-sided [26.14 to 31.41], Standard Error of Mean 1.48

17. Secondary Outcome: Change From Baseline in Urinary Hypoxanthine Levels at Day 1, Day 7, and Day 14
Description: Change from baseline in urinary hypoxanthine cumulative amounts at Day 1, Day 7 and Day 14
Time Frame: Baseline, Day 1, Day 7 and Day 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Number analyzed (Participants) | 7 | 3 | 11 | 9
mg
  Baseline (n=7,3,11,9) | 5.999 (2.4371) | 7.732 (1.5422) | 5.416 (2.3568) | 5.500 (1.9022)
  Change at Day 1 (n=7,3,11,9) | 2.435 (2.1850) [0.94 to 3.93] | 3.051 (2.5346) [0.76 to 5.34] | 1.600 (3.2414) | 1.486 (2.1230) [-0.08 to 3.16]
  Change at Day 7 (n=7,2,0,6) | 3.295 (3.1395) [1.80 to 4.79] | 8.714 (0.2294) [5.40 to 10.83] | NA (NA) [NA to NA] — No data due to cohort termination after 2 days of dosing. | 0.384 (0.9645) [-1.23 to 2.00]
  Change at Day 14 (n=6,2,0,6) | 4.291 (3.2263) [2.88 to 6.05] | 10.536 (0.9138) [7.22 to 12.66] | NA (NA) [NA to NA] — No data due to cohort termination after 2 days of dosing. | 0.870 (0.8776) [-0.75 to 2.49]
Statistical Analysis 1: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 0.90, 90% CI 2-sided [-1.31 to 3.10], Standard Error of Mean 1.29
Statistical Analysis 2: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 7; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 2.91, 90% CI 2-sided [0.71 to 5.11], Standard Error of Mean 1.29
Statistical Analysis 3: Comparison: Cohort 1: PF-06743649 2.5 mg to 10 mg vs Cohort 1 and 2: Placebo; Day 14; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 3.59, 90% CI 2-sided [1.33 to 5.85], Standard Error of Mean 1.33
Statistical Analysis 4: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 1; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 1.51, 90% CI 2-sided [-1.29 to 4.31], Standard Error of Mean 1.64
Statistical Analysis 5: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 7; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 7.73, 90% CI 2-sided [4.57 to 10.89], Standard Error of Mean 1.86
Statistical Analysis 6: Comparison: Cohort 1: PF-06743649 40 mg vs Cohort 1 and 2: Placebo; Day 14; Test type: Superiority or Other; Mixed Models Analysis; LS Mean Difference = 9.07, 90% CI 2-sided [5.91 to 12.23], Standard Error of Mean 1.86

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another, or 1 participant may have experienced both an AE and SAE during the study. All treated participants were included in the analysis.
Arm/Group | Cohort 1: PF-06743649 2.5 mg to 10 mg | Cohort 1: PF-06743649 40 mg | Cohort 2: PF-06743649 5 mg | Cohort 1 and 2: Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3 | 1/11 | 0/9
Other Adverse Events (participants affected / at risk) | 2/7 | 3/3 | 2/11 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-06743649 2.5 mg to 10 mg (N=7) | Cohort 1: PF-06743649 40 mg (N=3) | Cohort 2: PF-06743649 5 mg (N=11) | Cohort 1 and 2: Placebo (N=9)
Renal injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-06743649 2.5 mg to 10 mg (N=7) | Cohort 1: PF-06743649 40 mg (N=3) | Cohort 2: PF-06743649 5 mg (N=11) | Cohort 1 and 2: Placebo (N=9)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 1
Cystatin C increased (Investigations) | 0 | 3 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.